CLINICAL TRIAL: NCT00944892
Title: A Randomized,Double Blind,Placebo-controlled,Parallel Group,Repeat Dose Study of the Safety and Efficacy of REGN475 in Patients With Osteoarthritis of the Knee
Brief Title: A Study of the Safety and Efficacy of REGN475(SAR164877) in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R475-PN-0901
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Dose 1 (Experimental)
  Interventions: Drug: REGN475
- Dose 2 (Experimental)
  Interventions: Drug: REGN475
- Dose 3 (Experimental)
  Interventions: Drug: REGN475
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: REGN475 — 2 Administrations of REGN475 within 24 weeks.
  Arms: Dose 1; Dose 2; Dose 3
Other: Placebo — Placebo to match REGN475 doses
  Arms: Placebo

SUMMARY:
This is a double-blind, prospective, randomized study in which patients will be randomized to 1 of 4 treatment arms (3 active and 1 placebo).

Each patient will receive two doses of active medication or placebo, with study drug administered intravenously (IV). The primary goal of the study is to assess the safety and tolerability of repeat administrations of REGN475 compared to placebo in patients with osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 40 and ≤ 75 years of age.
2. Diagnosis of OA of the knee according to American College of Rheumatology (ACR) criteria, and experiencing moderate to severe pain in the index knee for at least 3 months prior to the screening visit.
3. Kellgren-Lawrence grade 2-3 radiographic severity of the index knee at or within 6 months prior to Screening.

Exclusion Criteria:

1. Significant concomitant illness including, but not limited to, cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease that would adversely affect the patient's participation in the study.
2. Patients with joint replacement in the affected knee.
3. Patients with peripheral neuropathy due to any reason.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The incidence of TEAEs in patients treated with REGN475 or placebo, reported between administration of study drug on Day 1 and the completion of study at the end of week 24 (Day 169). | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in The Western Ontario and McMaster Osteoarthritis Index (WOMAC) (total score as well as all 3 subscales: pain, stiffness and function). | 24 weeks
Patient assessment of response to treatment over time using the Patient Global Impression of Change. | 24 weeks
Change from baseline in patient-rated QOL using the Short-Form 12-Item Questionnaire (SF-12). | 24 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Anaheim, California
  - Tampa, Florida
  - Salt Lake City, Utah